CLINICAL TRIAL: NCT00894387
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Study to Evaluate the 6 Months Efficacy and Safety of Aliskiren Therapy on Top of Standard Therapy, on Morbidity and Mortality When Initiated Early After Hospitalization for Acute Decompensated Heart Failure
Brief Title: Six Months Efficacy and Safety of Aliskiren Therapy on Top of Standard Therapy, on Morbidity and Mortality in Patients With Acute Decompensated Heart Failure
Acronym: ASTRONAUT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPP100A2368; 2009-010236-18 (EudraCT Number)
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-10

CONDITIONS: Acute Decompensated Heart Failure; Congestive Heart Failure
Keywords: elevated BNP; reduced LVEF; Acute Heart Failure; Cardiovascular death; CHF; hospitalization; morbi-mortality trial; outcome study; endpoint driven; plasma renin activity; renin angiotensin; aldosterone system; direct renin inhibitors; BNP; KCCQ; eGFR
MeSH Terms: conditions — Heart Failure | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Aliskiren (Experimental): Randomized patients in this arm received, Aliskiren 150 mg once daily for 2 weeks. From week 2 upto 6 months , patients who could tolerate study medication were up-titrated to aliskiren 300 mg once daliy.
  Interventions: Drug: Aliskiren
- Placebo (Placebo Comparator): Randomized patients in this arm received matching placebo of Aliskiren. At week 2, Patients who could tolerate study medication were up-titrated to matching placebo of 300 mg aliskiren.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150 mg and Aliskiren 300 mg
  Other Names: Aliskiren®,; Tekturna®,; Rasilez®,; SPP100
  Arms: Aliskiren
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study evaluated the effect of early initiation of aliskiren therapy, compared to standard therapy, in the reduction of cardiovascular death and heart failure re-hospitalization events within 6 months, in congestive heart failure (CHF) patients hospitalized for an episode of acute decompensated heart failure.

ELIGIBILITY:
Inclusion criteria:

* Patient hospitalized with a primary diagnosis of worsening heart failure ≥ 18 years of age, male or female.
* Patients with a diagnosis of acute heart failure expressed by symptoms (dyspnea or fatigability - NYHA Class III-IV) and signs of fluid overload (i.e., jugular venous distension, edema or positive rales auscultation or pulmonary congestion on chest x-ray) at the time of hospitalization.

  * LVEF < 40% (measured within the last 6 months).
  * Hospitalization for ADHF and remain "stabilized" for at least 6 hours (defined as SBP ≥ 110 mm Hg after acute decompensated episode) and did not receive IV vasodilators (other than nitrates) and/or IV inotropic drugs at anytime from ADHF presentation to time of randomization.
* Elevated BNP at Visit 1 or at randomization (BNP ≥ 400 pg/ml).
* Patients with a history of chronic heart failure on standard therapy defined as requiring HF treatment for at least 30 days before the current hospitalization (NYHA Class II - IV).

Exclusion Criteria:

* Patients that required any use of IV vasodilators (except nitrates), and/or any IV inotropic therapy from the time of presentation for worsening HF to randomization.
* Concomitant use of ACEI and ARB at randomization.
* Right heart failure due to pulmonary disease.
* Diagnosis of postpartum cardiomyopathy.
* Myocardial infarction or cardiac surgery, including percutaneous transluminal coronary angioplasty (PTCA), within past 3 months.
* Patients with a history of heart transplant or who are on a transplant list.
* Unstable angina or coronary artery disease likely to require coronary artery bypass graft (CABG) or PTCA before randomization.

Other protocol-defined inclusion/exclusion criteria applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1639 (Actual)
Dates: Start 2009-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Study Director — Novartis
Locations (239):
- United States (32):
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Sylmar, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Hartford, Connecticut
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Macon, Georgia
  - Novartis Investigative Site, Oakbrook Terrace, Illinois
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, Lafayette, Louisiana
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Cherry Hill, New Jersey
  - Novartis Investigative Site, Newark, New Jersey
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Saratoga Springs, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Springfield, Tennessee
  - Novartis Investigative Site, Brownsville, Texas
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, Richmond, Virginia
- Argentina (9):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, San Nicolás de los Arroyos, Buenos Aires
  - Novartis Investigative Site, Corrientes, Corrientes Province
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Posadas, Misiones Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Santa Fe, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Quilmes
- Belgium (10):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Huy
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Mechelen
  - Novartis Investigative Site, Mol
  - Novartis Investigative Site, Namur
- Brazil (7):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Londrina, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (5):
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Colombia (6):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogotá, Cundinamarca
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cali
  - Novartis Investigative Site, Florida Blanca
- Czechia (8):
  - Novartis Investigative Site, Brno-Bohunice, Czech Republic
  - Novartis Investigative Site, Slaný, Czech Republic
  - Novartis Investigative Site, Znojmo, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Teplice
- Finland (2):
  - Novartis Investigative Site, Jyväskylä
  - Novartis Investigative Site, Turku
- France (7):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Le Chesnay
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Pontoise
  - Novartis Investigative Site, Toulouse
- Germany (34):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Bevensen
  - Novartis Investigative Site, Bad Nauheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bischofswerda
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Cloppenburg
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Cottbus
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Detmold
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Herrsching am Ammersee
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Konstanz
  - Novartis Investigative Site, Langen
  - Novartis Investigative Site, Ludwigslust
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Merseburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Nordhorn
  - Novartis Investigative Site, Paderborn
  - Novartis Investigative Site, Quedlinburg
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Sömmerda
  - Novartis Investigative Site, Weiden
- Hungary (7):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Balatonfüred
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Hódmezővásárhely
  - Novartis Investigative Site, Nagykanizsa
  - Novartis Investigative Site, Szolnok
  - Novartis Investigative Site, Zalaegerszeg
- India (13):
  - Novartis Investigative Site, Secunderabad, Andhra Pradesh
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, New Delhi, India
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Indore, M.p.
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Bangalore
  - Novartis Investigative Site, Hyderabad
- Israel (7):
  - Novartis Investigative Site, Nazareth, Israel
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Hadera
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Safed
  - Novartis Investigative Site, Tel Aviv
- Italy (25):
  - Novartis Investigative Site, Pavia, (pv)
  - Novartis Investigative Site, Verona, (vr)
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Lagosanto, FE
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Grosseto, GR
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Casarano, LE
  - Novartis Investigative Site, Lecce, LE
  - Novartis Investigative Site, Scorrano, LE
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Legnano, MI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Albano Laziale, RM
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Rimini, RN
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Legnago, VR
- Philippines (3):
  - Novartis Investigative Site, Quezon City, National Capital Region
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon City
- Poland (13):
  - Novartis Investigative Site, Krakow, Poland
  - Novartis Investigative Site, Grodzisk Wielkopolski
  - Novartis Investigative Site, Kłodzko
  - Novartis Investigative Site, Lódz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Ruda Śląska
  - Novartis Investigative Site, Swidnica
  - Novartis Investigative Site, Szczecin
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wałbrzych
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Zabrze
  - Novartis Investigative Site, Zamość
- Romania (5):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Târgovişte
  - Novartis Investigative Site, Timișoara
- Russia (7):
  - Novartis Investigative Site, Lyubertsy
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, S.-Petersburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Yaroslavl
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Slovakia (11):
  - Novartis Investigative Site, Liptovský Mikuláš, Slovak Republic
  - Novartis Investigative Site, Prešov, Slovak Republic
  - Novartis Investigative Site, Komárno, Slovakia
  - Novartis Investigative Site, Levice, Slovakia
  - Novartis Investigative Site, Nitra, Slovakia
  - Novartis Investigative Site, Trnava, Slovakia
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Kosice-Saca
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Lučenec
  - Novartis Investigative Site, Martin
- Spain (9):
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Villamartín, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Majadanonda, Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Valencia, Valencia
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
- Taiwan (6):
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Keelung
  - Novartis Investigative Site, Lin-Ko
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (10):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Istanbul, Turkey
  - Novartis Investigative Site, Atakum / Samsun
  - Novartis Investigative Site, Etlik / Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Kırıkkale
  - Novartis Investigative Site, Sivas
  - Novartis Investigative Site, Talas / Kayseri

REFERENCES:
- [Derived] Vaduganathan M, Cheema B, Cleveland E, Sankar K, Subacius H, Fonarow GC, Solomon SD, Lewis EF, Greene SJ, Maggioni AP, Bohm M, Zannad F, Butler J, Gheorghiade M. Plasma renin activity, response to aliskiren, and clinical outcomes in patients hospitalized for heart failure: the ASTRONAUT trial. Eur J Heart Fail. 2018 Apr;20(4):677-686. doi: 10.1002/ejhf.973. Epub 2017 Nov 16. PMID 29143416
- [Derived] Greene SJ, Butler J, Fonarow GC, Subacius HP, Ambrosy AP, Vaduganathan M, Triggiani M, Solomon SD, Lewis EF, Maggioni AP, Bohm M, Chioncel O, Nodari S, Senni M, Zannad F, Gheorghiade M; ASTRONAUT Investigators and Coordinators. Pre-discharge and early post-discharge troponin elevation among patients hospitalized for heart failure with reduced ejection fraction: findings from the ASTRONAUT trial. Eur J Heart Fail. 2018 Feb;20(2):281-291. doi: 10.1002/ejhf.1019. Epub 2017 Oct 17. PMID 29044915
- [Derived] Lund LH, Trochu JN, Meyns B, Caliskan K, Shaw S, Schmitto JD, Schibilsky D, Damme L, Heatley J, Gustafsson F. Screening for heart transplantation and left ventricular assist system: results from the ScrEEning for advanced Heart Failure treatment (SEE-HF) study. Eur J Heart Fail. 2018 Jan;20(1):152-160. doi: 10.1002/ejhf.975. Epub 2017 Sep 27. PMID 28960673
- [Derived] Gheorghiade M, Bohm M, Greene SJ, Fonarow GC, Lewis EF, Zannad F, Solomon SD, Baschiera F, Botha J, Hua TA, Gimpelewicz CR, Jaumont X, Lesogor A, Maggioni AP; ASTRONAUT Investigators and Coordinators. Effect of aliskiren on postdischarge mortality and heart failure readmissions among patients hospitalized for heart failure: the ASTRONAUT randomized trial. JAMA. 2013 Mar 20;309(11):1125-35. doi: 10.1001/jama.2013.1954. PMID 23478743
- [Derived] Gheorghiade M, Albaghdadi M, Zannad F, Fonarow GC, Bohm M, Gimpelewicz C, Botha J, Moores S, Lewis EF, Rattunde H, Maggioni A; ASTRONAUT investigators and study coordinators. Rationale and design of the multicentre, randomized, double-blind, placebo-controlled Aliskiren Trial on Acute Heart Failure Outcomes (ASTRONAUT). Eur J Heart Fail. 2011 Jan;13(1):100-6. doi: 10.1093/eurjhf/hfq209. Epub 2010 Nov 30. PMID 21123186

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 2134 screened patients (including
  1 patient who was screened twice), 1639 patients were randomized.
Period: Overall Study
Arm/Group | Aliskiren | Placebo
Started | 821 ("Started" indicates all randomized patients) | 818
Safety Set | 808 | 810
Full Analysis Set | 808 | 807
Completed Primary Efficacy Phase (6 m) | 717 | 707
Completed Secondary Efficacy Phase (12m) | 654 | 640
Completed | 646 ("Completed" indicates patients whose treatment duration completed as per protocol) | 643
Not Completed | 175 | 175
Not completed — Adverse Event | 44 | 45
Not completed — Abnormal Laboratory values | 2 | 2
Not completed — Unsatisfactory therapeutic effect | 0 | 1
Not completed — Lost to Follow-up | 3 | 5
Not completed — Administrative problems | 2 | 2
Not completed — Death | 77 | 76
Not completed — Protocol Deviation | 4 | 0
Not completed — Patient's request | 25 | 30
Not completed — Other (Missing) | 5 | 3
Not completed — Mis-randomized | 13 | 9
Not completed — GCP non-compliance | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Placebo | Total
Number analyzed (Participants) | 808 | 807 | 1615
Age Continuous [Mean (Standard Deviation); unit: years] | 64.7 (12.44) | 64.5 (11.88) | 64.6 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 197 | 368
  Male | 637 | 610 | 1247

OUTCOME MEASURES:

1. Secondary Outcome: Time to Event Analysis: Number of Patients Experienced the First Confirmed Occurrence of Either Cardiovascular Death or Heart Failure (HF) Re-hospitalization Within 12 Months
Description: Time to first confirmed occurrence of either cardiovascular death or heart failure re-hospitalization within 12 months of randomization was the key secondary efficacy variable. For the primary efficacy analysis, an event will be considered for the analysis if it occurs on or before Day 395 (394 days from randomization). The secondary composite endpoint is the the composite of cardiovascular death or heart faliure re-hospitalization within 12 months.
Time Frame: 12 months
Population: Full analysis set (FAS) consisted of randomized patients who had received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 808 | 807
Participants
  Secondary Composite Endpoint | 283 | 301
  Cardiovascular death | 126 | 137
  Heart faliure re-hospitalization | 212 | 224

2. Secondary Outcome: Change From Baseline in the Clinical Summary Score to 1 Month, 6 Months and 12 Months
Description: Symptom reduction and reduction in physical limitations was assessed using the clinical summary score of the Kansas City Cardiomyopathy Questionnaire (KCCQ). The KCCQ is a self-administered questionnaire and contains 23 items, covering physical function, clinical symptoms, social function, self-efficacy and knowledge, and Health-Related Quality of Life (QoL), including limitations, frequency, bother, change in condition, understanding, levels of enjoyment and satisfaction. Each scale score was calculated as the mean of its item scores and transformed to a 0-100 scale, with higher score indicating higher level of functioning. A score of 100 represents perfect health whereas a score of 0 represents death. A positive change in score from baseline indicates an improvement.
Time Frame: Baseline, 1 months, 6 months and 12 months
Population: Full analysis set included all randomized patients who had taken at least one dose of drug. 'n' in each category indicates patients with assessable data both at baseline and corresponding time points.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 808 | 807
units on a scale
  1 Month (n= 574, 571) | 24.13 (0.903) | 23.58 (0.908)
  6 Months (n= 485, 474) | 26.54 (1.004) | 24.51 (1.016)
  12 Months (n= 241, 230) | 24.82 (1.268) | 24.70 (1.291)

3. Secondary Outcome: Time to Event Analysis: Number of Patients With First Cardiovascular (CV) Event Hospitalized for an Acute Heart Faliure (AHF) Event Within 6 Months
Description: A cardiovascular event defined as CV death, heart faliure re-hospitalization, non-fatal myocardial infarction (MI), nonfatal stroke, sudden death with resuscitation.
Time Frame: 6 months
Population: Full analysis set included all randomized patients who had taken at least one dose of drug.
Measure: Number; unit: Participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 808 | 807
Participants
  Cardiovascular event | 209 | 233
  Cardiovascular death | 77 | 85
  Heart faliure re-hospitalization | 153 | 166
  All-cause myocardial infarction | 14 | 23
  Fatal myocardial infarction | 2 | 6
  Non-fatal myocardial infarction | 12 | 22
  All-cause stroke | 13 | 22
  Fatal stroke | 6 | 4
  Non-fatal stroke | 13 | 22
  Resuscitated sudden death | 3 | 8

4. Secondary Outcome: Time to Event Analysis: Number of Patients With All-cause Mortality Hospitalized for an AHF Event Within 12 Months
Time Frame: 12 months
Population: Full ananlysis set included all randomized patients who had at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 808 | 807
Participants | 144 | 148

5. Primary Outcome: Time to Event Analysis: Number of Patients Experienced the First Confirmed Occurrence of Either Cardiovascular Death or Heart Failure (HF) Re-hospitalization Within 6 Months
Description: Time to first confirmed occurrence of either cardiovascular death or heart failure re-hospitalization within 6 months of randomization was the primary efficacy variable. For the primary efficacy analysis, an event will be considered for the analysis if it occurs on or before Day 190 (189 days from randomization). The primary composite endpoint is the the composite of cardiovascular death or heart faliure re-hospitalization within 6 months.
Time Frame: 6 months
Population: Full analysis set (FAS) consisted of randomized patients who had received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 808 | 807
Participants
  Primary Composite Endpoint | 201 | 214
  Cardiovascular death | 77 | 85
  Heart faliure re-hospitalization | 153 | 166

6. Secondary Outcome: Change From Baseline in N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) Level at 1 Month, 6 Months, and 12 Months
Description: The reported Least square means, and Confidential Interval were from a repeated measures model on log transformed NT-proBNP data containing treatment, visit, and region as factors, log baseline NT-proBNP as a continuous covariate and treatment by visit and visit by log baseline NT-proBNP as interaction terms.
Time Frame: Baseline, 1 month, 6 months and 12 months
Population: Full analysis set included all randomized patients who had taken at least one dose of study drug. 'n' in each category indicates patients with assessable date at baseline and each corresponding time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 808 | 807
pg/mL
  Month 1 (n= 669, 675) | 0.86 [0.81 to 0.91] | 0.95 [0.90 to 1.00]
  Month 6 (n= 569, 556) | 0.64 [0.59 to 0.70] | 0.76 [0.70 to 0.82]
  Month 12 (n=447, 425) | 0.62 [0.56 to 0.68] | 0.74 [0.67 to 0.82]

7. Secondary Outcome: Time to Event Analysis: Number of Patients With First Cardiovascular (CV) Event Hospitalized for an Acute Heart Faliure (AHF) Event Within 12 Months
Description: as for outcome 3
Time Frame: 12 months
Population: Full analysis set included all randomized patients who had taken at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 808 | 807
Participants
  Cardiovascular event | 293 | 321
  Cardiovascular death | 126 | 137
  Heart faliure re-hospitalization | 212 | 224
  All-cause myocardial infarction | 18 | 38
  Fatal myocardial infarction | 4 | 12
  Non-fatal myocardial infarction | 16 | 36
  All-cause stroke | 18 | 27
  Fatal stroke | 6 | 7
  Non-fatal stroke | 18 | 27
  Resuscitated sudden death | 5 | 10

ADVERSE EVENTS:
Arm/Group | Aliskiren | Placebo
Serious Adverse Events (participants affected / at risk) | 421/808 | 435/810
Other Adverse Events (participants affected / at risk) | 367/808 | 333/810
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren (N=808) | Placebo (N=810)
Anaemia (Blood and lymphatic system disorders) | 6 | 5
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 | 0
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Jaundice acholuric (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 3 | 3
Acute left ventricular failure (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 9 | 15
Angina pectoris (Cardiac disorders) | 9 | 10
Angina unstable (Cardiac disorders) | 7 | 6
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 3 | 3
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Arteriospasm coronary (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 14 | 16
Atrial flutter (Cardiac disorders) | 3 | 2
Atrial tachycardia (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 2 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 11 | 14
Cardiac failure (Cardiac disorders) | 147 | 155
Cardiac failure acute (Cardiac disorders) | 58 | 60
Cardiac failure chronic (Cardiac disorders) | 50 | 62
Cardiac failure congestive (Cardiac disorders) | 21 | 31
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 7 | 3
Cardiogenic shock (Cardiac disorders) | 7 | 6
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 2 | 1
Cardiorenal syndrome (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 2 | 2
Coronary artery disease (Cardiac disorders) | 4 | 2
Heart valve incompetence (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Low cardiac output syndrome (Cardiac disorders) | 1 | 0
Myocardial fibrosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 11 | 11
Myocardial ischaemia (Cardiac disorders) | 3 | 3
Palpitations (Cardiac disorders) | 2 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 2
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 3 | 1
Ventricular arrhythmia (Cardiac disorders) | 2 | 4
Ventricular dysfunction (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 4 | 5
Ventricular tachycardia (Cardiac disorders) | 10 | 6
Vertigo (Ear and labyrinth disorders) | 4 | 2
Cataract (Eye disorders) | 3 | 0
Eye haemorrhage (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 1
Retinal detachment (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 4
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 5
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 8 | 3
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2
Asthenia (General disorders) | 1 | 3
Cardiac death (General disorders) | 3 | 3
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 6 | 0
Death (General disorders) | 21 | 25
Device breakage (General disorders) | 0 | 1
Device lead issue (General disorders) | 1 | 0
Device malfunction (General disorders) | 1 | 4
Drug intolerance (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 4
General physical health deterioration (General disorders) | 2 | 3
Generalised oedema (General disorders) | 2 | 2
Implant site haematoma (General disorders) | 0 | 1
Medical device complication (General disorders) | 0 | 1
Metaplasia (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 3
Necrosis (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 7 | 1
Oedema peripheral (General disorders) | 3 | 6
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Soft tissue inflammation (General disorders) | 1 | 0
Stent malfunction (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 5 | 7
Sudden death (General disorders) | 9 | 5
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1
Heart transplant rejection (Immune system disorders) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Arthritis infective (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 6 | 6
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 3 | 4
Cellulitis (Infections and infestations) | 1 | 3
Citrobacter sepsis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 4
Endocarditis (Infections and infestations) | 0 | 3
Erysipelas (Infections and infestations) | 2 | 1
Gangrene (Infections and infestations) | 2 | 3
Gastroenteritis (Infections and infestations) | 2 | 3
Gastroenteritis norovirus (Infections and infestations) | 1 | 1
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 2
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 2
Lung infection pseudomonal (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 2
Osteomyelitis acute (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 25 | 27
Pneumonia legionella (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 2
Pseudomembranous colitis (Infections and infestations) | 2 | 0
Pseudomonas bronchitis (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 3 | 2
Sepsis (Infections and infestations) | 8 | 5
Septic shock (Infections and infestations) | 5 | 5
Skin infection (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 1
Subacute endocarditis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 4 | 5
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Wound infection pseudomonas (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Dermatitis artefacta (Injury, poisoning and procedural complications) | 1 | 0
Electric shock (Injury, poisoning and procedural complications) | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 4 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Optic nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 2
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Anticoagulation drug level above therapeutic (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 3 | 1
Blood osmolarity decreased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Coagulation test abnormal (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 2 | 1
Renal function test abnormal (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 0 | 3
Weight increased (Investigations) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid intake reduced (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 12 | 12
Hyperosmolar state (Metabolism and nutrition disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 7 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 5
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatobiliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anterior spinal artery syndrome (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 9 | 15
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Diabetic hyperglycaemic coma (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 2 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 3
Hypokinesia (Nervous system disorders) | 1 | 1
Intracranial haematoma (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 5 | 9
Loss of consciousness (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0
Myasthenia gravis crisis (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 3 | 4
Sensory disturbance (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 2 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 11 | 13
Transient ischaemic attack (Nervous system disorders) | 0 | 3
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
Uraemic encephalopathy (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 1
Screaming (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 1
Anuria (Renal and urinary disorders) | 0 | 1
Bladder tamponade (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal artery thrombosis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 6 | 8
Renal failure acute (Renal and urinary disorders) | 20 | 12
Renal failure chronic (Renal and urinary disorders) | 1 | 3
Renal impairment (Renal and urinary disorders) | 5 | 4
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 18
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Gastric bypass (Surgical and medical procedures) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 1
Extremity necrosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 3
Hypertensive crisis (Vascular disorders) | 1 | 3
Hypertensive emergency (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 24 | 16
Intra-abdominal haematoma (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 2
Peripheral ischaemia (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 2 | 1
Phlebitis (Vascular disorders) | 1 | 0
Venous haemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren (N=808) | Placebo (N=810)
Diarrhoea (Gastrointestinal disorders) | 49 | 36
Hyperkalaemia (Metabolism and nutrition disorders) | 155 | 128
Hypokalaemia (Metabolism and nutrition disorders) | 42 | 53
Dizziness (Nervous system disorders) | 35 | 43
Renal impairment (Renal and urinary disorders) | 47 | 33
Cough (Respiratory, thoracic and mediastinal disorders) | 59 | 53
Hypotension (Vascular disorders) | 117 | 83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.